CLINICAL TRIAL: NCT01364870
Title: Effect of TENS on Hyperalgesia, Pain With Movement, and Function After TKR
Brief Title: Effect of TENS for Pain and Function After Total Knee Replacement
Acronym: TANK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara A Rakel (Other)
Responsible Party: Sponsor-Investigator, Barbara A Rakel, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200706725
Record Dates: First submitted 2011-05-31; First posted 2011-06-03 (Estimated); Results first posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-10

CONDITIONS: Unilateral Primary Osteoarthritis of Knee; Primary Osteoarthritis of Knee Nos
Keywords: Knee OA; TENS; Total knee replacement; Knee arthroplasty; total unilateral knee replacement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Active TENS (Active Comparator): High-frequency intense TENS provided with the EMPI Select TENS. The generator emits a balanced, asymmetrical, biphasic waveform and has buttons for variation of frequency and amplitude. A rate modulation frequency of 50pps and 150pps every 0.5 seconds will be used with a pulse width of 150 microseconds (μs).
  Interventions: Device: Active TENS
- Placebo TENS (Placebo Comparator): Subjects randomized to the placebo group will use an EMPI TENS Select device that emits a current for 45 seconds then shuts off. They will be asked when they first feel the current, then the device will be turned down a half-point to provide "treatment" at a sub-sensory level. This unit displays an active indicator light suggesting to the subject that the unit is actively emitting current. At discharge, subject will be sent home with an adequate supply of batteries and asked to change batteries when the device goes below 4 bars, further suggesting that the device is actively working.
  Interventions: Device: Placebo TENS
- Standard Care (No Intervention): Subjects randomized to "Standard Care" will be given no TENS unit.

INTERVENTIONS:
Device: Placebo TENS — Subjects randomized to the placebo group will use an EMPI TENS Select device that emits a current for 45 seconds then shuts off. They will be asked when they first feel the current, then the device will be turned down a half-point to provide "treatment" at a sub-sensory level. This unit displays an active indicator light suggesting to the subject that the unit is actively emitting current. At discharge, subject will be sent home with an adequate supply of batteries and asked to change batteries when the device goes below 4 bars, further suggesting that the device is actively working.
  Arms: Placebo TENS
Device: Active TENS — High-frequency intense TENS provided with the EMPI Select TENS. The generator emits a balanced, asymmetrical, biphasic waveform and has buttons for variation of frequency and amplitude. A rate modulation frequency of 50pps and 150pps every 0.5 seconds will be used with a pulse width of 150 microseconds (μs).
  Arms: Active TENS

SUMMARY:
Our primary hypothesis is that TENS decreases pain with movement by reducing hyperalgesia. Minimizing the severe pain experienced during required activities in the immediate postoperative period will promote functional recovery and prevent the development of new chronic pain syndromes.

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis of the knee
* Speak English
* Unilateral total knee replacement

Exclusion Criteria:

* No ambulation, assisted or otherwise
* Use of TENS by subject in past 5 yrs
* Current use of TENS by someone else in subject's household
* Stroke or other condition which seriously impairs sensation in legs or ability to follow directions.
* Condition that precludes use of TENS (pacemaker, allergy to nickel, etc.)
* Chronic pain (other than in surgical knee) that is currently being treated or is severe. (Do not exclude for fibromyalgia).

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2008-05; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Rakel, PhD, RN, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

REFERENCES:
- [Derived] Dindo L, Zimmerman MB, Hadlandsmyth K, StMarie B, Embree J, Marchman J, Tripp-Reimer T, Rakel B. Acceptance and Commitment Therapy for Prevention of Chronic Postsurgical Pain and Opioid Use in At-Risk Veterans: A Pilot Randomized Controlled Study. J Pain. 2018 Oct;19(10):1211-1221. doi: 10.1016/j.jpain.2018.04.016. Epub 2018 May 17. PMID 29777950

RESULTS

PARTICIPANT FLOW:
Groups:
- Intense TENS: High-frequency intense TENS provided with the EMPI Select TENS. The generator emits a balanced, asymmetrical, biphasic waveform and has buttons for variation of frequency and amplitude. A rate modulation frequency of 50pps and 150pps every 0.5 seconds will be used with a pulse width of 150 microseconds (μs).
  Intense TENS (EMPI Select TENS): High-frequency intense TENS provided with the EMPI Select TENS. The generator emits a balanced, asymmetrical, biphasic waveform and has buttons for variation of frequency and amplitude. A rate modulation frequency of 50pps and 150pps every 0.5 seconds will be used with a pulse width of 150 microseconds (μs).
Period: Overall Study
Arm/Group | Intense TENS | Placebo TENS | Standard Care
Started | 122 | 123 | 72
Completed | 100 | 93 | 58
Not Completed | 22 | 30 | 14
Not completed — Withdrawal by Subject | 13 | 24 | 10
Not completed — Adverse Event | 8 | 6 | 4
Not completed — Protocol Violation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intense TENS | Placebo TENS | Standard Care | Total
Number analyzed (Participants) | 122 | 123 | 72 | 317
Age, Continuous [Mean (Full Range); unit: Years] | 62.7 [41 to 90] | 61.9 [40 to 82] | 62.2 [42 to 86] | 62.3 [40 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 65 | 42 | 172
  Male | 57 | 58 | 30 | 145
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 118 | 121 | 71 | 310
  Unknown or Not Reported | 3 | 1 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 114 | 117 | 68 | 299
  More than one race | 2 | 2 | 1 | 5
  Unknown or Not Reported | 6 | 4 | 3 | 13
Pain with knee range of motion: Extension [Mean (Full Range); unit: scores on a scale] — While subject's knee extension is measured, they report their pain on 0-20 Numeric Rating Scale (where 0 is "no pain" and 20 is "pain as bad as you can imagine").
  scores on a scale | 6.69 [0 to 20] | 7.03 [0 to 20] | 8.03 [0 to 20] | 7.13 [0 to 20]
Pain with walking [Mean (Full Range); unit: scores on a scale] — While subject was walking, they report their pain on 0-20 Numeric Rating Scale (where 0 is "no pain" and 20 is "pain as bad as you can imagine").
  scores on a scale | 6.1 [0 to 20] | 6.29 [0 to 20] | 7.65 [0 to 20] | 6.52 [0 to 20]
Pain at rest [Mean (Full Range); unit: scores on a scale] — While subject is sitting and not moving, they report their pain on 0-20 Numeric Rating Scale (where 0 is "no pain" and 20 is "pain as bad as you can imagine").
  scores on a scale | 2.92 [0 to 15] | 3.35 [0 to 18] | 3.76 [0 to 19] | 3.28 [0 to 19]
Pressure Pain Threshold [Mean (Full Range); unit: kilopascal (kPa)] | 264.08 [51 to 853.3] | 251.02 [36.3 to 770] | 247 [28 to 681.5] | 255.16 [28 to 853.3]
Heat Pain Threshold [Mean (Full Range); unit: Degrees Celsius] | 43.3 [35.7 to 49.6] | 43.3 [35.8 to 49.8] | 43.6 [35.8 to 48] | 43.4 [35.7 to 49.8]
Heat Pain Tolerance [Mean (Full Range); unit: Degrees Celsius] | 47.4 [42.5 to 52] | 46.8 [35.9 to 50] | 47.1 [38.3 to 51] | 47.1 [35.9 to 52]
Knee Range of Motion: Extension [Mean (Full Range); unit: Degrees] | -5 [-30 to 10] | -4.8 [-24 to 8] | -6.5 [-26 to 4] | -5.3 [-30 to 10]
Gait Speed Test [Mean (Full Range); unit: feet in 15 seconds] | 61.9 [8.8 to 117] | 62.7 [13.8 to 120] | 60.5 [15.4 to 122.5] | 61.9 [8.8 to 122.5]
Range of motion: Flextion [Mean (Full Range); unit: Degrees] | 112.5 [61 to 140] | 115.4 [35 to 140] | 109.8 [58 to 142] | 113 [35 to 142]

OUTCOME MEASURES:

1. Primary Outcome: Self-Reported Pain With Movement
Description: While subject's knee extension is measured, they report their pain on 0-20 Numeric Rating Scale (where 0 is "no pain" and 20 is "pain as bad as you can imagine").
Time Frame: 1 day post-op
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Intense TENS | Placebo TENS | Standard Care
Number analyzed (Participants) | 111 | 121 | 68
scores on a scale | 9.5 [0 to 20] | 10 [0 to 20] | 14 [0 to 20]
Statistical Analysis 1: Comparison: Intense TENS vs Placebo TENS vs Standard Care; There were instances of missing data due to patient time restraints and patient refusal; Test type: Superiority; p = 0.016, Kruskal-Wallis — The p value was adjusted using Bonferroni's method to account for the multiple comparisons

2. Primary Outcome: Self-reported Pain With Walking (From Iowa Gait Test)
Description: Subjects are instructed to walk as quickly as they safely can for 15 seconds. Their pain was assessed with a Numeric Rating Scale (where 0 is "no pain" and 20 is "pain as bad as you can imagine").
Time Frame: 2 days post-op
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Intense TENS | Placebo TENS | Standard Care
Number analyzed (Participants) | 105 | 115 | 67
scores on a scale | 8 [0 to 20] | 10 [0 to 20] | 10 [0 to 20]
Statistical Analysis 1: Comparison: Intense TENS vs Placebo TENS vs Standard Care; There were instances of missing data due to patient time restraints and patient refusal; Test type: Superiority; p = 0.008, Kruskal-Wallis — P-value was adjusted using Bonferroni's method to account for multiple comparisons

ADVERSE EVENTS:
Arm/Group | Intense TENS | Placebo TENS | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/122 | 0/123 | 0/72
Serious Adverse Events (participants affected / at risk) | 7/122 | 3/123 | 6/72
Other Adverse Events (participants affected / at risk) | 4/122 | 7/123 | 2/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intense TENS (N=122) | Placebo TENS (N=123) | Standard Care (N=72)
Blood clot in non-surgical leg (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Blood clot in surgical leg (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Infection in surgical knee (Infections and infestations) | 4 (4) | 2 (2) | 3 (3)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Readmission to hospital for medication adjustment (General disorders) | 1 (1) | 0 (0) | 1 (1)
Surgery to remove broken drain tube (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Injury (torn hamstring) during physical therapy (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intense TENS (N=122) | Placebo TENS (N=123) | Standard Care (N=72)
Fall at home (Injury, poisoning and procedural complications) | 4 (4) | 7 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No